CLINICAL TRIAL: NCT06610773
Title: Effectiveness and Safety of Human Umbilical Cord Mesenchymal Stem Cells for the Treatment of HPV High-risk Infection
Brief Title: HUC-MSC for Treatment of High-risk HPV Infection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2024(CR)-001; HX-2021-007 (Other Grant/Funding Number: Shanghai Shanghai East Hospital)
Record Dates: First submitted 2024-08-28; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Human Papillomavirus Viruses; Mesenchymal Stem Cells
Keywords: HPV; hUC-MSC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental group (Experimental): 1×10^6/Kg UC-MSCs (resuspended in 100 mL normal saline containing 5% albumin) are infused intravenously to the high-risk HPV persistant infected patients at a controlled rate of 60-80 drops/min
  Interventions: Biological: hUC-MSCs
- Control group (Placebo Comparator): Normal saline containing 5% albumins are infused intravenously with an equal volume, similar suspension and appearance package as UC-MSCs to the high-risk HPV persistant infected patients at a controlled rate of 60-80 drops/min
  Interventions: Biological: Saline+albumin

INTERVENTIONS:
Biological: hUC-MSCs — 1×10^6/Kg hUC-MSCs (suspended in 100 mL normal saline containing 5% albumin) are infused intravenously to patients at a controlled rate of 60-80 drops/min.
  Other Names: Umbilical Cord Mesenchymal Stem Cells
  Arms: Experimental group
Biological: Saline+albumin — Normal saline containing 5% albumin had a similar suspension and appearance package to hUC-MSCs, but no MSCs
  Arms: Control group

SUMMARY:
To evaluate the safety and initial effectiveness of human umbilical cord mesenchymal stem cells in HPV clearance.

DETAILED DESCRIPTION:
Cervical cancer is one of the most common malignant tumors of the female reproductive system with the highest incidence. Nearly 99.7% of cervical cancer is caused by HPV infection. Studies have shown that the persistent infection of high-risk human papillomavirus (HR-HPV) is an independent risk factor for cervical cancer which can lead to a 250-fold increased risk of high-grade cervical intraepithelial neoplasia (CIN). In patients with persistent HR-HPV infection for more than 12 months, the risk of diagnosis of high-grade squamous intraepithelial lesions of the cervix by 30 months increased to 21%. In the process of progression from HPV infection to cervical cancer, cervical precancerous lesions, namely intraepithelial neoplasia (CIN), will be experienced. Therefore, effective control of HPV infection, especially the elimination of persistent HR-HPV infection, will greatly reduce the incidence of CIN and cervical cancer. It is an urgent clinical need to actively intervene in patients with persistent infections for more than one year with a clinical significance at present.

Mesenchymal Stem Cells (MSCs) are a class of pluripotent stem cells derived from the mesoderm and ectoderm of early development, which can be easily obtained from a variety of tissue organs, having a strong proliferation and multidirectional differentiation potential in vitro. hUC-MSCs have a great effect on immune regulation and anti-inflammatory properties with a fewer ethical, availability, safety issues and a broader prospect in clinical research and application. At present, many experimental data have proved that MSCs can enhance the clearance of virus by immune cells in vivo, and have a certain application prospect in fighting virus infection. The purpose of this study was to evaluate the safety and therapeutic efficacy of human umbilical cord mesenchymal stem cells (HUC-MSCs) in clearing HPV infection, and to provide clinical basis for HUC-MSCs to clear HPV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 25-60 with a sexual history of more than 2 years;
2. Confirmed HPV infection by HPV-24 test;Patients diagnosed with high-risk human papillomavirus (HR-HPV) persistent infection; (note: the HR HPV: HPV 16/18/31/33/35/39/45/51/52/53/56/58/59/66/68; 15 types)
3. The subjects were not participating in other clinical trials at the same time, and had no other anti-HPV drugs or intervention therapy recently;
4. If the pregnancy test is negative and the subjects have fertility potential, they agree to use effective contraception during the study period and within 6 months of completion or termination of the study;
5. Voluntarily participate in and agree to cooperate in accordance with the requirements of the program, and sign the informed consent.

Exclusion Criteria:

1. Women who are preparing for pregnancy, pregnancy or breastfeeding;
2. Pathological diagnosis of high-grade squamous intraepithelial lesion (HSIL) or cervical cancer;
3. Previous HPV vaccinations;
4. A history of severe drug allergies, or allergies to stem cell products or other biologics;
5. Previous cervical site physical therapy or related surgical history;
6. Patients with severe immune dysfunction (such as AIDS, systemic lupus erythematosus and other immune system diseases or history of organ transplantation, malignant tumor chemotherapy history), serious cardiovascular, liver, kidney, nervous, hematopoietic system diseases or malignant tumors, or mental diseases;
7. Recent use of other antiviral drugs, immunosuppressants, immunomodulators or steroid hormones that affect the immune system;
8. Patients with acute genital tract inflammation or pelvic inflammation;
9. Those who have participated in or are participating in clinical trials of other drugs within three months;
10. Other conditions considered inappropriate by the investigator for inclusion in this clinical trial.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events-The incidence rate of allergic reaction | 1day,1st,4th,12th,and 36th week
  The allergic reaction rate on the 1st day, 1st week, 4th week, 12th week, and 36th week after the infusion.
The 24 type HPV viral load | -28th~0day,4th,12th,and 36th week
  HPV24 genotypes test is classified from female genitourinary secretions and exfoliating cells of cervix by fluorescent PCR before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 4th week, 12th week, and 36th week after the infusion.

SECONDARY OUTCOMES:
The percentage of CD3+ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the percentage（%）of CD3+ before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week, 12th and 36th week after the infusion.
The percentage of CD4+ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the percentage（%）of CD4+ before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week, 12th and 36th week after the infusion.
The percentage of CD8+ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the percentage（%） of CD8 before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week, 12th and 36th week after the infusion.
The percentage of CD19+ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the percentage（%）of CD19+ before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week, 12th and 36th week after the infusion
The percentage of CD16+/CD56+ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the percentage（%） of CD16+/CD56+ before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week, 12th and 36th week after the infusion.
The serum level of IFN-γ | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the level of IFN-γ (pg/mL) before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 12th week, and 36th week after the infusion.
The serum level of IL-6 | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the level of IL-6 (pg/mL) before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week,12th week, and 36th week after the infusion.
The serum level of IL-8 | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the level of IL-8 (pg/mL) before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week,12th week, and 36th week after the infusion.
The serum level of IL-10 | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the level of IL-10 (pg/mL) before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 4th week,12th week, and 36th week after the infusion.
The serum level of TNF-α | -28th~0day,1day,1st,4th,12th,and 36th week
  The peripheral blood serum of the patients will be collected to detect the level of TNF-α (pg/mL) before the infusion of hUC-MSCs (Any day from 28th to 1st day) and on the 1st day, 1st week, 12th week, and 36th week after the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, M.D,.PH.D., Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Shanghai Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No